CLINICAL TRIAL: NCT02007733
Title: Assessment of Severe Dehydration in Children With Diarrhea in Bangladesh
Brief Title: DeHydration: Assessing Kids Accurately
Acronym: DHAKA
Status: Completed | Type: Observational
Sponsor: Rhode Island Hospital (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: 470125; 1K01TW009208-01A1 (NIH)
Record Dates: First submitted 2013-11-25; First posted 2013-12-11 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2015-10

CONDITIONS: Severe Dehydration
Keywords: Diarrhea; Dehydration; Children; Resuscitation; Clinical Prediction Rule; Low Income Country; Bangladesh
MeSH Terms: conditions — Dehydration; Diarrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Derivation Cohort: The derivation cohort includes patients enrolled in the first phase of the study, from February 2014 to June 2014. All children enrolled in this study will receive the same interventions, which include collection of regular weights to establish percent weight change with rehydration, clinical assessment of dehydration status, and ultrasound of the IVC and aorta.
  Interventions: Other: Serial Weights; Other: IVC/Aorta Ultrasound; Other: Clinical Assessment
- Validation Cohort: The validation cohort includes patients enrolled in the second phase of the study, from March 2015 to May 2015. All children enrolled in this study will receive the same interventions, which include collection of regular weights to establish percent weight change with rehydration, clinical assessment of dehydration status, and ultrasound of the IVC and aorta.
  Interventions: Other: Serial Weights; Other: Clinical Assessment

INTERVENTIONS:
Other: Serial Weights — We will collect serial weights on all children enrolled in this study.
Other: IVC/Aorta Ultrasound — We will perform an ultrasound assessment of the IVC and Aorta size in each child enrolled.
  Groups: Derivation Cohort
Other: Clinical Assessment — We will perform a clinical assessment of dehydration status in each child enrolled in the study, as well as collect data on mid-upper arm circumference, length, symptoms and demographic information.

SUMMARY:
Diarrhea is the second leading cause of death in children worldwide, and accurately assessing dehydration status remains a crucial step in preventing morbidity and mortality from this disease. While children with severe dehydration require immediate treatment with intravenous fluids, children with mild to moderate dehydration have a significant reduction in hospital length of stay and fewer adverse events when treated with relatively inexpensive oral rehydration solution (ORS). While several clinical scales have been developed for assessing dehydration in children, these scales have never been prospectively validated in a low-income country setting, where the vast majority of diarrhea morbidity and mortality occurs in children.

The investigators hypothesize that new clinical and ultrasound-based tools will improve the diagnosis of severe dehydration in children with diarrhea in low-income countries, reducing the morbidity and mortality that occurs as a result of under-diagnosis of severe dehydration as well as the adverse events and inappropriate utilization of scarce resources that occurs as a result of over-diagnosis of severe dehydration.

DETAILED DESCRIPTION:
Background:

Children under five experience 1.7 billion episodes of diarrhea each year, resulting in 36 million cases of severe disease and 700,000 deaths, or 10% of all child deaths worldwide. As the severity of diarrheal disease can vary quite widely in children, accurately assessing dehydration status remains a crucial step in preventing morbidity and mortality. While children with severe dehydration require immediate treatment with intravenous fluids to prevent hemodynamic compromise, organ ischemia, and death, children with mild to moderate dehydration have a significant reduction in hospital length of stay and fewer adverse events when treated with relatively inexpensive oral rehydration solution (ORS). The World Health Organization (WHO), the US Centers for Disease Control and Prevention (CDC), and the European Society of Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) recommend separating children with acute diarrhea into three groups to determine management based on the presence or absence of various clinical signs: no dehydration (<3%), some dehydration (3-9%), and severe dehydration (>9%). These authorities recommend treating children with some dehydration with ORS and limiting IV hydration to children with severe dehydration, in order to prevent the inappropriate utilization of scarce hospital resources and the adverse events associated with a more liberal use of IV hydration in children. However, no clinical prediction model for severe dehydration has ever been empirically derived and validated in a developing world setting, where the vast majority of diarrheal deaths occur in children each year.

Study Objectives:

As part of this study, the investigators will derive a new clinical prediction rule for severe dehydration in children with diarrhea in the developing world. In addition, the investigators will validate and assess the reliability of ultrasound of the inferior vena cava (IVC) for predicting severe dehydration in children with diarrhea. Finally, the investigators will compare the accuracy of each of these new diagnostic tools to that of the WHO scale, the current standard for assessing dehydration in most low-income countries.

Study Design:

The investigators will enroll a prospective cohort of children under five admitted with diarrhea and dehydration to the Dhaka Hospital of the International Center for Diarrheal Disease Research, Bangladesh (ICDDR,B). Research staff will identify eligible children on arrival and obtain informed consent from their guardian. Children will be weighed on arrival and assessed clinically for the presence or absence of signs of dehydration. A brief ultrasound of the IVC will also be performed. Children will then be rehydrated according to standard hospital protocols, with their weight checked regularly until they achieve a stable, post-hydration weight. Greater than 9% difference between admission weight and stable weight (or post-illness weight) will be considered the gold standard for severe dehydration, against which the investigators will determine the accuracy of our new clinical and ultrasound-based assessment tools.

Ethical Protection of Human Subjects:

Children enrolled are very unlikely to be exposed to any additional risks or discomforts, either mental or physical, as a result of participating in this study. Study procedures will include physical exam and ultrasound, neither of which will expose children to increased harm, and study procedures will not delay any immediately necessary care, such as IV fluids. All data collected will be kept strictly confidential in a password-protected database. In addition to obtaining ethical approval from the Lifespan Institutional Review Board (IRB), the investigators have also already obtained approval from the ICDDR,B Ethical Review Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 years (60 months) or younger
2. History of diarrhoea (defined as 3 or more loose stools per day)
3. Children observed in the rehydration ward

Exclusion Criteria:

1. Chronic diarrhoea (greater than 2 week duration)
2. Clear alternative diagnosis to gastroenteritis on presentation
3. Previously enroled in this research study

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under five with acute diarrhea observed in the rehydration ward of the Dhaka Hospital of ICDDR,B.
Sampling Method: Probability Sample
Enrollment: 1396 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver-Operator Characteristic (ROC) curve for predictors of severe diarrheal disease | 2 weeks
  We will follow all enrolled children for up to a maximum of 2 weeks to assess the percent change between initial dehydrated weight and stable rehydration weight or post-illness weight. Greater than 9% weight change or death prior to achieving stable weight will be our criterion standard for severe disease. We will then determine the area under the Receiver-Operator Characteristic (ROC) curves for our newly derived clinical scale (DHAKA scale); for ultrasound of the IVC to Aorta ratio; and for the WHO scale as predictors of severe diarrheal disease in children enrolled in our study.

SECONDARY OUTCOMES:
Area under the receiver operating curve for predictors of some dehydration | 2 weeks
  We will follow all enrolled children for up to a maximum of 2 weeks to assess the percent change between initial dehydrated weight and stable rehydration weight or post-illness weight. 3-9% weight change between arrival and stable weight or post-illness weight will be our criterion standard for some dehydration. We will then determine the area under the Receiver-Operator Characteristic (ROC) curves for our newly derived clinical scale (DHAKA scale); for ultrasound of the IVC to Aorta ratio; and for the WHO scale as predictors of some dehydration in children enrolled in our study.

OTHER OUTCOMES:
Sub-group analyses | 2 weeks
  We will perform subgroup analyses for all of our predictors of dehydration in children by age, nutrition status, and type of diarrhea (watery versus bloody).

CONTACTS AND LOCATIONS:
Overall Officials: Adam C. Levine, MD, MPH, Principal Investigator — Brown University
Locations (1):
- Dhaka Hospital of ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Result] Levine AC, Glavis-Bloom J, Modi P, Nasrin S, Rege S, Chu C, Schmid CH, Alam NH. Empirically Derived Dehydration Scoring and Decision Tree Models for Children With Diarrhea: Assessment and Internal Validation in a Prospective Cohort Study in Dhaka, Bangladesh. Glob Health Sci Pract. 2015 Aug 18;3(3):405-18. doi: 10.9745/GHSP-D-15-00097. PMID 26374802
- [Result] Levine AC, Glavis-Bloom J, Modi P, Nasrin S, Atika B, Rege S, Robertson S, Schmid CH, Alam NH. External validation of the DHAKA score and comparison with the current IMCI algorithm for the assessment of dehydration in children with diarrhoea: a prospective cohort study. Lancet Glob Health. 2016 Oct;4(10):e744-51. doi: 10.1016/S2214-109X(16)30150-4. Epub 2016 Aug 23. PMID 27567350
- [Derived] Modi P, Nasrin S, Hawes M, Glavis-Bloom J, Alam NH, Hossain MI, Levine AC. Midupper Arm Circumference Outperforms Weight-Based Measures of Nutritional Status in Children with Diarrhea. J Nutr. 2015 Jul;145(7):1582-7. doi: 10.3945/jn.114.209718. Epub 2015 May 13. PMID 25972523
- See also: Principal Investigator Website — https://research.brown.edu/myresearch/Adam_Levine